CLINICAL TRIAL: NCT03021460
Title: Phase I Study of Pembrolizumab in Combination With Ibrutinib in the Treatment of Unresectable or Metastatic Melanoma
Brief Title: Pembrolizumab and Ibrutinib in Treating Patients With Stage III-IV Melanoma That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1577; NCI-2017-00079 (Registry Identifier: CTRP (Clinical Trials Reporting Program)); 16-002462 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — ibrutinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ibrutinib, pembrolizumab) (Experimental): Patients receive ibrutinib PO daily on days 1-28 of cycle 1 and days 1-21 of cycle 2 and subsequent cycles. Patients also receive pembrolizumab IV over 30 minutes on day 8 of cycle 1 and day 1 of cycle 2 and subsequent cycles. Cycle 1 continues for 28 days and subsequent cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial studies the best dose of ibrutinib when given together with pembrolizumab in treating patients with stage III-IV melanoma that cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Ibrutinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and ibrutinib may work better in treating patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of ibrutinib in combination with pembrolizumab in patients with advanced melanoma. (Phase I) II. To estimate the overall response rate treated at the maximum tolerated dose of ibrutinib in combination with pembrolizumab in patients with advanced melanoma. (Dose expansion cohort)

SECONDARY OBJECTIVES:

I. To assess the safety and adverse-event profiles of combination of ibrutinib with pembrolizumab in patients with advanced melanoma.

II. To evaluate the overall response rate (ORR) in patients advanced melanoma receiving ibrutinib and pembrolizumab.

III. To evaluate the duration of response, progression-free survival (PFS), and overall survival (OS) in patients with advanced melanoma receiving ibrutinib and pembrolizumab.

IV. To assess the effect of treatment with ibrutinib and pembrolizumab on Th1/Th2 immune polarity.

EXPLORATORY OBJECTIVES:

I. To assess the CD8 T cell response to multiple melanoma-associated antigens, and to correlate CD8 T cell responses with changes in Th1/Th2 immune polarity.

II. To assess changes in plasma cytokines induced by treatment with ibrutinib and pembrolizumab.

III. To assess the change in potential biomarkers, such as tumor-bound and soluble PD-L1 levels and tumor-infiltrating lymphocytes, that may correlate with treatment responses.

OUTLINE: This is a dose-escalation study of ibrutinib.

Patients receive ibrutinib orally (PO) daily on days 1-28 of cycle 1 and days 1-21 of cycle 2 and subsequent cycles. Patients also receive pembrolizumab intravenously (IV) over 30 minutes on day 8 of cycle 1 and day 1 of cycle 2 and subsequent cycles. Cycle 1 continues for 28 days and subsequent cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION- INCLUSION CRITERIA
* Diagnosis of unresectable stage III or metastatic melanoma (stage IV) not amenable to local therapy
* At least one non-nodal lesion considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (that is, a lesion whose longest diameter can be accurately measured as >= 1.0 cm with computed tomography [CT] scan, CT component of a positron emission tomography [PET]/CT, or magnetic resonance imaging [MRI]) or at least one malignant lymph node is considered measurable by RECIST criteria (that is, its short axis is >= 1.5 cm when assessed by CT scan)

  * NOTE: tumor lesions in a previously irradiated area are not considered measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Provide informed written consent
* Patient is willing to undergo treatment and monitoring at the enrolling institution
* Willing to provide tissue and blood samples for correlative research purposes
* REGISTRATION- INCLUSION CRITERIA
* Histologic or cytologic confirmation of unresectable stage III or metastatic melanoma (stage IV) not amenable to local therapy
* Only if patient has had previous exposure to anti-PD-1 or anti-PD-L1 therapy:

  * Patient had disease progression on or within 6 months after anti-PD-1/anti-PD-L1 therapy in the metastatic setting OR
  * Patient had disease progression within 6 months after the last dose of adjuvant/neoadjuvant anti-PD-1/anti-PD-L1 treatment
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration)

  * Criteria must be met without a transfusion =< four weeks prior to registration
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 X upper limit of normal (ULN); if total bilirubin > 1.5 X ULN then direct bilirubin =< ULN (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (aspartate transaminase [AST]) and alanine aminotransferase (alanine transaminase [ALT]) =< 2.5 x ULN OR =< 5 X ULN for patients with liver metastases (obtained =< 14 days prior to registration)
* Creatinine =< 1.5 X ULN and creatinine clearance (CrCL) >= 30 ml/min per Cockcroft Gault formula (obtained =< 14 days prior to registration)
* Patients of childbearing potential only, negative urine pregnancy test done =< 7 days prior to study registration

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study medication; adequate contraception is defined as 2 methods of birth control (e.g., hormonal contraceptives, intrauterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide) or prior surgical sterilization, or abstinence from heterosexual activity
* Prior treatment with ibrutinib or prior exposure to BTK inhibitors
* Uveal melanoma
* Current use of warfarin or other vitamin K antagonists
* Require continuous treatment with a strong CYP3A inhibitor
* Currently participating or has participated in a study of an investigational cancer therapy agent or using an investigational device within 28 days prior to study registration
* Live vaccines within 28 days prior to study pre-registration
* Invasive surgical procedure within 28 days prior to study pre-registration
* History of clinically severe (e.g., requires chronic immunosuppressive therapy, [e.g., cyclosporine A, tacrolimus]) autoimmune disease (e.g., ulcerative colitis, lupus), or history of organ transplant
* Known history of human immunodeficiency virus (HIV) infection, active infection with hepatitis B virus or hepatitis C virus, or any uncontrolled active systemic infection
* Gastrointestinal disease that might inhibit ibrutinib absorption (e.g., malabsorption syndrome, resection of the stomach or a large portion of small bowel, or partial/complete bowel obstruction), or unable to swallow capsules
* Active central nervous system metastases and/or carcinomatous meningitis

  * Note: Patients with untreated brain metastasis will be excluded; patients with previously treated brain metastases may participate provided they meet the following criteria:

    * Inactive (without evidence of progression which is documented by CT or MRI within 90 days prior to registration), AND
    * On =< 10 mg/day prednisone or equivalent for at least 28 days prior pre-registration
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Clinically significant cardiovascular disease such as unstable angina, myocardial infarction, or acute coronary syndrome within =< 180 days prior to registration, symptomatic or uncontrolled arrhythmia, congestive heart failure, or any class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Other active malignancy =< 3 years prior to pre-registration; note: if there is a history of prior malignancy, the patient must not be receiving other specific treatment for cancer

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome =< 6 months prior to pre-randomization
* Known bleeding disorders (von Willebrand's disease or hemophilia)
* History of ischemic stroke or intracranial hemorrhage =< 180 days prior to pre-registration
* Currently active, clinically significant hepatic impairment Child-Pugh class A, B or C according to the Child Pugh classification
* Unresolved toxicities from prior anti-cancer therapy, defined as not resolved to Common Terminology Criteria for Adverse Events (CTCAE, version [v]4.0) grade 0 or 1, or to the levels dictated in the inclusion/exclusion criteria with the exceptions of alopecia and peripheral neuropathy
* REGISTRATION- EXCLUSION
* Failure to confirm histologically or cytologically unresectable stage III or metastatic melanoma (stage IV) not amenable to local therapy
* Prior chemotherapy, immunotherapy, radioactive, or biological cancer therapy (including monoclonal antibody [mAb]) =< 28 days prior to registration
* Received a strong cytochrome P450 (CYP) 3A inhibitor =< 7 days prior to registration
* Concurrent systemic immunosuppressant therapy =< 21 days prior to registration
* Recent infection requiring systemic antibiotic treatment that was completed =< 14 prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (Phase I) | Up to start of second course of treatment
  Will be defined as the highest dose level among those tested where at most one out of 6 patients develops a dose limiting toxicity prior to the start of their second course of treatment. The maximum grade of each type of toxicity will be recorded for each patient. For each toxicity reported by dose level, the percentage of patients developing any degree of that toxicity as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.
Tumor response (dose expansion cohort) | Up to 5 years
  Estimates of tumor response and binomial confidence intervals will be reported.

SECONDARY OUTCOMES:
Tumor response evaluated according to Response Evaluation Criteria in Solid criteria (RECIST) | Up to 5 years
  A patient whose tumor has met the RECIST criteria for complete response or partial response on two consecutive evaluations at least 8 weeks apart is considered to have had a tumor response.
Progression-free survival | From study entry to the documentation of disease progression, assessed up to 5 years
  Will be examined in an exploratory and hypothesis-generating fashion.
Overall survival | From study entry to death due to any cause, assessed up to 5 years
  Will be examined in an exploratory and hypothesis-generating fashion.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Yao Y, Yan Y, Suman VJ, Dietz AB, Erskine CL, Dimou A, Markovic SN, McWilliams RR, Montane HN, Block MS. Phase I study of pembrolizumab in combination with ibrutinib for the treatment of unresectable or metastatic melanoma. Front Immunol. 2025 Feb 4;16:1491448. doi: 10.3389/fimmu.2025.1491448. eCollection 2025. PMID 39967670
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials